CLINICAL TRIAL: NCT06935708
Title: Intrathecal Morphine Versus Thoracic Epidural Analgesia for Open Colorectal Cancer Surgery: a Randomized Controlled Trial
Brief Title: Intrathecal Morphine Versus Epidural Analgesia for Open Colon Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Meri Mirceta (Other)
Responsible Party: Sponsor-Investigator, Meri Mirceta, Anesthesiologist, Doctor of Medicine (MD), University Hospital of Split
Organization: University Hospital of Split (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2181-147/01/06/LJ.Z.-25-02
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Carcinoma; Analgesia, Postoperative; Laparotomy
Keywords: postoperative pain; analgesia; epidural; intrathecal morphine; laparotomy
MeSH Terms: conditions — Colorectal Neoplasms; Agnosia; Pain, Postoperative | interventions — Analgesia, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural group (Active Comparator): Epidural group will have an epidural catheter inserted in the T10/11 or T11/12 interspace using a midline approach. The epidural space will be identified by a loss of resistance to saline with a Tuohy 18G epidural needle. Subsequently, the epidural catheter will be inserted 4-6 cm into the epidural space and a test-dose of 2% lidocaine, 50 mg, to detect intrathecal misplacement will be given. Epidural group will subsequently receive intraoperative intermittent epidural analgesia followed by postoperative continuous infusion of a levobupivacaine and fentanyl mixture.
  Interventions: Procedure: Epidural Analgesia
- Spinal group (Experimental): In Spinal group, 25 G or 27 G pencil point needle, depending on the preference of the anesthesiologist, will be inserted at L2-L3 or L3-L4 intervertebral space and 300 μg of preservative-free morphine (Morphine Kalceks ®, Kalceks, AS, Riga, Latvija, 10mg/ml) diluted with sterile saline to a volume of 3 mL will be injected intrathecally.
  Interventions: Drug: Intrathecal Morphine

INTERVENTIONS:
Drug: Intrathecal Morphine — In Spinal group, 25 G or 27 G pencil point needle, depending on the preference of the anesthesiologist, will be inserted at L2-L3 or L3-L4 intervertebral space and 300 μg of preservative-free morphine (Morphine Kalceks ®, Kalceks, AS, Riga, Latvija, 10mg/ml) diluted with sterile saline to a volume of 3 mL will be injected intrathecally.
  Arms: Spinal group
Procedure: Epidural Analgesia — Epidural analgesia with levobupivacaine and fentanyl mixture. For intraoperative intermittent analgesia, Epidural group will be given a loading dose of 5-10 milliliters of a mixture of 10 micrograms per milliliter (μg/mL) of fentanyl (Fentanyl Piramal Critical Care, 50 mcg/ml) and 0.25% levobupivacaine (Levobupivakain Kabi 5 mg/ml), followed by intermittent 4-5 mL boluses as needed throughout the surgery. Postoperative continuous epidural analgesia in the epidural group will consist of 2 μg/mL fentanyl added to 0.1 % levobupivacaine at the rate 5-8 mL/h during the first 24 hours after surgery.
  Arms: Epidural group

SUMMARY:
Effective pain management after abdominal surgery is essential for recovery. This study compares two pain relief methods-intrathecal morphine (a single spinal injection) and continuous epidural analgesia-for patients undergoing open colorectal cancer surgery.

The investigators expect intrathecal morphine to provide equal pain relief at rest 24 hours after surgery, while epidural analgesia may be more effective during movement. By 48 to 72 hours, both methods should offer similar pain control. The epidural group may require fewer additional pain medications but could experience more side effects, including a higher risk of low blood pressure and technical difficulties. Additionally, these patients may have a slightly longer hospital stay. In contrast, the intrathecal morphine group may have fewer overall side effects. Despite these differences, patient satisfaction, sleep quality, and recovery are expected to be similar in both groups.

By evaluating these methods, this study aims to determine the most effective and safe approach to post-surgical pain management, improving comfort and recovery outcomes for patients.

DETAILED DESCRIPTION:
Participants of this study will be randomly selected adult patients with colorectal carcinoma undergoing open colorectal resection who fulfill the inclusion criteria and sign the informed consent for participation.

This sample represents the population of adult patients with colorectal cancer undergoing open surgery by ERAS protocol in a tertiary hospital of a high-developed country.

Patients will be randomly divided into Epidural group (E group) or Spinal group (S group) and will receive different intraoperative and postoperative analgesia plans.

E group will be treated as a control group. Patients in S group will receive intrathecal morphine as analgesia for colorectal resection and it will be treated as experimental group.

Anesthesia induction and maintenance will be the same in both groups. The primary outcome is pain intensity at rest measured with the Numeric Rating Scale (0 = no pain and 10 = worst pain) 24 hours after surgery. Secondary outcome measures are analgesic consumption, time to rescue analgesia, patient satisfaction, quality of sleep, length of hospital stay, time to return of bowel function, and adverse events (such as respiratory depression, nausea or vomiting, hypotension and bradycardia).

Postoperative continuous epidural analgesia in the E group will consist of 2 μg/mL fentanyl added to 0.1 % levobupivacaine at the rate 5-8 mL/h during the first 24 hours after surgery.

Additional epidural boluses will be allowed by the nursing staff for pain Numerical Rating Scale (NRS)≥4.

Both groups will receive standard multimodal analgesic protocol with the goal of postoperative pain NRS<4: intravenous (iv) paracetamol 1 g up to 4 times per day and iv metamizole 2.5 g up to 2 times per day and tramadol 50-100 mg iv as needed. In the control group, epidural analgesia will be used for postoperative pain relief for up to 24 h. An algorithm of postoperative rescue analgesia is established for each group.

Rescue antiemetics will be given in case of postoperative nausea and vomiting (PONV): metoclopramide 10 mg iv up to 3 times per day and granisetron 1 mg iv up to 3 times per day.

Severe pruritus will be treated with antihistamines or naloxone 40 mcg iv.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with colorectal carcinoma undergoing laparoscopic abdominal surgery aged 18-80 years, ASA classification I-III, Body Mass Index (BMI) 15-35 kg/m2.

Exclusion Criteria:

* abnormal coagulation function, defined as prothrombin time or activated partial prothrombin time above standard laboratory values or an international normalised ratio (INR) ≥1.4; or receiving ongoing therapeutic anticoagulation,
* thrombocytopenia, defined as a platelet count <80×10 9 L-1,
* pre-existing skin infection at the neuraxial anesthesia puncture site,
* pre-existing neurologic deficit, including peripheral neuropathy,
* patients with dementia or other medical condition that includes communication difficulties,
* patients with bradycardia (pulse <50/min) or with conduction block (2nd or 3rd degree)
* history of opioid abuse,
* allergies to any of the drugs used in the study.

Additionally, patients converted from laparoscopy to laparotomy due to technical surgical issues, patients with postoperative surgical complications (need for revision) or if epidural catheter placement/spinal anesthesia is unsuccessful even after an attempt by a senior anesthesiologist will also be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Pain intensity at rest 24 hours after surgery. | 24 hours
  Level of pain intensity will be validated using Numeric Rating Scale ranging from 0-10.

SECONDARY OUTCOMES:
Pain scores at rest and during movement at 1, 3, 6, 48, and 72 hours, and during movement at 24 h after surgery | 1, 3, 6, 24, 48, and 72 hours after surgery
  Numeric Rating Scale
Intraoperative use of fentanyl. | For the duration of surgery.
  Total amount of administered fentanyl in mg.
Time to the first request for rescue analgesia. | From the time of the surgery until the time to the first request for rescue analgesia (up to 3 days after the surgery)
  Measured in minutes.
Consumption of tramadol and metamizole. | Total amount of tramadol and metamizole within 72 hours after surgery.
  Measured in mg.
Patient satisfaction | 24, 48, and 72 hours after surgery
  Measured with a 5-point Likert scale.
Quality of sleep. | 24, 48, and 72 hours after surgery
  Measured with a 5-point Likert scale.
Quality of Recovery | 72 hours after surgery
  Measured with a 15-item Quality of Recovery 15 (QoR-15) scale.
Length of stay (LOS) in HDU (high dependency unit) | From the time of the admission to HDU until ward discharge (up to 30 days)
  Time to ward discharge in hours.
Length of hospital stay | Form the day of surgery until hospital discharge (up to 90 days)
  Time from surgery to hospital discharge in days.
Time to ambulation | From the end of surgery until patient ambulation (up to 30 days)
  Measured in hours, defined as the patient independently getting out of bed.
Time to gastro-intestinal recovery | From the end of surgery until the first documented stool, flatus or oral intake (up to 3 days)
  First stool or flatus after surgery measured in hours, time to oral intake
Sedation score | After extubation and 24 hours after surgery.
  Measured with a Ramsay sedation scale (1-6)
Incidence of respiratory depression | Within 24 hours after surgery.
  Respiratory rate <8 /min or need for assisted ventilation.
Incidence of nausea or vomiting | Within 24 hours after surgery.
Incidence of shivering, pruritus, hypotension, bradycardia. | Within 24 hours after surgery
  Hypotension defined as systolic blood pressure less than 90 mmHg or diastolic less than 50 mmHg, mean arterial pressure < 60 mmHg, or decline >20% from baseline, and bradycardia defined as heart rate <50/min.
Incidence of post-dural puncture headache | Within 72 hours after surgery.
Incidence of technique failure | Perioperative
  Need to convert to a second analgesic technique due to multiple reasons, e.g., inability to perform spinal puncture, inability to insert an epidural catheter, inadequate analgesia, epidural catheter malfunction, or dislodgement.
Postoperative complications | Until hospital discharge (up to 90 days)
  Postoperative complications will be classified according to the Clavien Dindo Classification (1, 2, 3 a, 3 b, 4 a, 4 b, 5).
Readmission rate | Within 30 days after surgery
  Readmission is defined as patient admission related to surgical procedure within 30 days after initial discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: No